CLINICAL TRIAL: NCT05625412
Title: A Phase 1, Open-label, Multicenter Study of BMS-986360/CC-90001 Alone and in Combination With Chemotherapy or Nivolumab in Advanced Solid Tumors
Brief Title: A Study of BMS-986360/CC-90001 Alone and in Combination With Chemotherapy or Nivolumab in Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IM043-004; 2022-500930-27 (EudraCT Number)
Record Dates: First submitted 2022-11-15; First posted 2022-11-22 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Advanced Solid Tumors
Keywords: Solid tumors; Nivolumab; Chemotherapy; BMS-986360; CC-90001
MeSH Terms: interventions — CC-90001; Docetaxel; Nivolumab; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- BMS-986360 (Experimental)
  Interventions: Drug: BMS-986360
- BMS-986360 + Docetaxel (Experimental)
  Interventions: Drug: BMS-986360; Drug: Docetaxel
- BMS-986360 + Nivolumab (Experimental)
  Interventions: Drug: BMS-986360; Drug: Nivolumab
- BMS-986360 + Capecitabine (Experimental)
  Interventions: Drug: BMS-986360; Drug: Capecitabine

INTERVENTIONS:
Drug: BMS-986360 — Specified dose on specified days
  Other Names: CC-90001
Drug: Docetaxel — Specified dose on specified days
  Other Names: Taxotere®
  Arms: BMS-986360 + Docetaxel
Drug: Nivolumab — Specified dose on specified days
  Other Names: Opdivo®; BMS-936558
  Arms: BMS-986360 + Nivolumab
Drug: Capecitabine — Specified dose on specified days
  Other Names: Xeloda®
  Arms: BMS-986360 + Capecitabine

SUMMARY:
The aim of this study is to assess the safety and tolerability of BMS-986360 as monotherapy and in combination with chemotherapy or nivolumab in participants with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Participants in Part 1 must have histologic or cytologic confirmation of non-small cell lung cancer (NSCLC), metastatic triple negative breast cancer (mTNBC), squamous cell carcinoma of head and neck (SCCHN), pancreatic adenocarcinoma (PAAD), renal cell carcinoma (RCC), microsatellite-stable colorectal carcinoma (MSS CRC), or sarcoma, that is advanced (metastatic, recurrent, and/or unresectable) with measurable disease per RECIST v1.1. In Part 2, only participants with histologic confirmation of advanced NSCLC or mTNBC with measurable disease per RECIST v1.1 are eligible.
* In Part 2, archival biopsy collected within 3 months of screening with no intervening therapy (formalin-fixed, paraffin embedded [FFPE] blocks or a minimum of 20 freshly cut unstained FFPE slides with an associated pathological report) or fresh biopsy collection at Screening and fresh biopsy collection at cycle 3 day 1 (C3D1) (± 5 days) are mandatory, while it is strongly encouraged but optional at progression. Therefore, the participant in Part 2 must have a suitable tumor lesion for the biopsy procedure, as judged by the investigator, in order to be eligible for the study.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.
* Participants resistant/refractory to or intolerant of existing standard therapies known to provide clinical benefit (in addition, participants with NSCLC must be resistant or refractory to anti-PD-(L)1-based immunotherapy)

Exclusion Criteria:

* Participants with primary central nervous system (CNS) disease, or tumors with CNS metastases as the only disease site, will be excluded. Participants with controlled brain metastases, however, will be allowed to enroll. Controlled brain metastases are defined as no radiographic progression for at least 4 weeks following radiation and/or surgical treatment (or 4 weeks of observation if no intervention is clinically indicated), no longer taking steroids for at least 2 weeks prior to first dose of study intervention, and with no new or progressive neurological signs and symptoms.
* Participants with a condition requiring systemic treatment with corticosteroids (> 10 mg daily prednisone equivalent) within 14 days or other immunosuppressive medications within 30 days of randomization. Inhaled or topical steroids and adrenal replacement steroid doses > 10 mg daily prednisone equivalent are permitted in the absence of active autoimmune disease.
* Participants with concurrent malignancy or history of prior malignancy active within 2 years (except history of early-stage basal/squamous cell skin cancer or non-invasive or in situ cancers who have undergone definitive treatment) are excluded unless treatment was completed at least 2 years before randomization and the participant has no evidence of disease.
* Participants with NSCLC with known or not tested for epidermal growth factor receptor (EGFR) or V-raf murine sarcoma viral oncogene homolog B1 (BRAF) V600E mutations, or anaplastic lymphoma kinase (ALK) or receptor tyrosine kinase (ROS1) translocations sensitive to available targeted inhibitor therapy

Other protocol-defined inclusion/exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2022-12-09 (Actual); Primary Completion 2025-05-12 (Actual); Study Completion 2025-05-12 (Actual)

PRIMARY OUTCOMES:
Number of participants with Adverse Events (AEs) | Up to approximately 2 years
Number of participants with Serious Adverse Events (SAEs) | Up to approximately 2 years
Number of participants with Dose-Limiting Toxicities (DLTs) | Up to approximately 2 years
Number of participants with AEs leading to discontinuation | Up to approximately 2 years
Number of deaths | Up to approximately 2 years

SECONDARY OUTCOMES:
Maximum observed plasma concentration (Cmax) | Up to approximately 2 years
Time of maximum observed plasma concentration (Tmax) | Up to approximately 2 years
Area under the plasma concentration-time curve (AUC) | Up to approximately 2 years
Part 1: Objective response rate (ORR) based on Response Evaluation Criteria in Solid Tumors (RECIST v1.1) by investigator | Up to approximately 2 years
Part 2: ORR based on RECIST v1.1 by blinded independent central review (BICR) assessment | Up to approximately 2 years
Part 1: Duration of Response (DOR) based on RECIST v1.1 by investigator | Up to approximately 2 years
Part 2: DOR based on RECIST v1.1 by BICR assessment | Up to approximately 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (35):
- United States (8):
  - Local Institution - 0029, Los Angeles, California
  - Local Institution - 0051, Los Angeles, California
  - Local Institution - 0026, New Orleans, Louisiana
  - Local Institution - 0001, Hackensack, New Jersey
  - Local Institution - 0018, Huntersville, North Carolina
  - Local Institution - 0028, Nashville, Tennessee
  - Local Institution - 0027, San Antonio, Texas
  - Local Institution - 0046, West Valley City, Utah
- Argentina (3):
  - Local Institution - 0033, Ciudad Autónoma de Buenos Aires, Buenos Aires
  - Local Institution - 0030, CABA, Buenos Aires F.D.
  - Local Institution - 0031, Buenos Aires
- Australia (4):
  - Local Institution - 0010, Darlinghurst, New South Wales
  - Local Institution - 0061, St Leonards, New South Wales
  - Local Institution - 0008, Brisbane, Queensland
  - Local Institution - 0063, Frankston, Victoria
- Canada (2):
  - Local Institution - 0003, Ottawa, Ontario
  - Local Institution - 0005, Toronto, Ontario
- Chile (3):
  - Local Institution - 0047, Santiago, Santiago Metropolitan
  - Local Institution - 0035, Santiago, Santiago Metropolitan
  - Local Institution - 0034, Santiago, Santiago Metropolitan
- France (4):
  - Local Institution - 0049, Marseille, Provence-Alpes-Côte d'Azur Region
  - Local Institution - 0052, Villejuif, Val-de-Marne
  - Local Institution - 0048, Paris
  - Local Institution - 0050, Toulouse
- Italy (3):
  - Local Institution - 0057, Rozzano, Milano
  - Local Institution - 0059, Candiolo, Torino
  - Local Institution - 0065, Padua
- Mexico (4):
  - Local Institution - 0041, Zapopan, Jalisco
  - Local Institution - 0038, Mexico City, Mexico City
  - Local Institution - 0039, Monterrey, Nuevo León
  - Local Institution - 0037, Puebla City
- Spain (4):
  - Local Institution - 0053, Barcelona, Catalunya [Cataluña]
  - Local Institution - 0055, Madrid, Madrid, Comunidad de
  - Local Institution - 0056, Madrid, Madrid, Comunidad de
  - Local Institution - 0064, Seville

IPD SHARING:
Plan to Share IPD: No
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myers Squibb's data sharing policy and process can be found at: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosurecommitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.BMSClinicalTrials.com